CLINICAL TRIAL: NCT04250051
Title: Phase 1 Trial of Ivosidenib and FLAG Chemotherapy in Relapsed/Refractory IDH1+ Acute Myeloid Leukemia (AML)
Brief Title: Ivosidenib and Combination Chemotherapy for the Treatment of IDH1 Mutant Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 19H05; STU00210558 (CTRP (Clinical Trial Reporting Program)); NU 19H05 (Other: Northwestern University); P30CA060553 (NIH); NCI-2019-08390 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Acute Myeloid Leukemia; Recurrent Myelodysplastic Syndrome; Recurrent Myeloproliferative Neoplasm; Refractory Acute Myeloid Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; fludarabine phosphate; ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (combination chemotherapy, ivosidenib) (Experimental): INDUCTION: Patients receive filgrastim SC QD on days 0-6, fludarabine phosphate IV QD over 30 minutes on days 1-5, cytarabine IV QD over 4 hours on days 1-5, and ivosidenib PO QD on days 7-28. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive filgrastim SC QD on days 0-5, fludarabine phosphate IV QD over 30 minutes on days 1-4, cytarabine IV QD over 4 hours on days 1-4, and ivosidenib PO QD on days 1-28. Treatment continues for 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive ivosidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Biological: Filgrastim; Drug: Fludarabine; Drug: Fludarabine Phosphate; Drug: Ivosidenib

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo

SUMMARY:
This phase I trial studies the side effects and best dose of ivosidenib when given together with combination chemotherapy for the treatment of 1DH1 mutant acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory). Ivosidenib may stop the growth of cancer cells by blocking the IDH1 mutation and some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fludarabine phosphate, cytarabine, and filgrastim, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ivosidenib with combination chemotherapy may work better in treating patients with acute myeloid leukemia compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of ivosidenib in combination with fludarabine, cytarabine, plus granulocyte-colony stimulating factor (G-CSF) (FLAG) chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of ivosidenib in combination with FLAG chemotherapy.

II. To determine the rate of complete remission (CR + complete remission with incomplete hematological recovery [CRi] + complete remission with incomplete platelet recovery [CRp]) with ivosidenib in combination with FLAG chemotherapy.

III. To evaluate the 1 year progression free survival. IV. To evaluate the 1 year overall survival. V. To assess the number of patients that receive allogeneic stem cell transplant after ivosidenib in combination with FLAG chemotherapy.

EXPLORATORY OBJECTIVES:

I. To assess for minimal residual disease negativity by polymerase chain reaction (PCR) for IDH1 mutations after treatment with ivosidenib in combination with FLAG chemotherapy.

II. To assess for minimal residual disease negativity by PCR for IDH1 mutations after 3 cycles of maintenance therapy.

OUTLINE:

INDUCTION: Patients receive filgrastim subcutaneously (SC) once daily (QD) on days 0-6, fludarabine phosphate intravenously (IV) QD over 30 minutes on days 1-5, cytarabine IV QD over 4 hours on days 1-5, and ivosidenib orally (PO) QD on days 7-28. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive filgrastim SC QD on days 0-5, fludarabine phosphate IV QD over 30 minutes on days 1-4, cytarabine IV QD over 4 hours on days 1-4, and ivosidenib PO QD on days 1-28. Treatment continues for 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive ivosidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every month for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed/refractory primary (ie, de novo) or secondary (progression of myelodysplastic syndrome [MDS] or myeloproliferative neoplasms [MPN], or therapy-related) acute myeloid leukemia (AML) according to the World Health Organization (WHO) classification with >= 5% leukemic blasts in the bone marrow
* Patients may have received prior therapies and there are no limits on number of therapies

  * Note: There is a requirement of 7 day washout from prior therapy or 5 half-lives, whichever is shorter
* Patient must have documentation of an IDH1 R132 mutation obtained prior to registration. IDH mutational status will be assessed locally
* Patients must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted
* Patient is willing and able to adhere to the study visit schedule and other protocol requirements
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal (ULN), unless considered due to leukemic organ involvement (within 28 days prior to registration)
* Serum total bilirubin < 1.5 x ULN (within 28 days prior to registration)

  * Higher levels are acceptable if these can be attributed to ineffective erythropoiesis, =< 3 times the upper limit of normal for Gilbert's syndrome (eg, a gene mutation in UGT1A1), or leukemic organ involvement
* Serum creatinine or creatinine clearance < 2 x ULN or >= 30 mL/min based on the Modification of Diet in Renal Disease (MDRD) glomerular filtration rate (GFR) (within 28 days prior to registration)
* Patients must agree to serial bone marrow aspirate/biopsies
* Females of childbearing potential (FOCBP) may participate, providing they meet the following conditions: Agree to practice true abstinence from sexual intercourse or to use two highly effective contraceptive methods, of which one must be a barrier method (eg, combined [containing estrogen and progestogen] or progestogen only associated with inhibition of ovulation, oral, injectable, intravaginal, patch, or implantable hormonal contraceptive; bilateral tubal occlusion; intra-uterine device; intrauterine hormone-releasing system; or male partner sterilization [note that a vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FOCBP trial participant and that a vasectomized partner has received medical assessment of the surgical success]) at screening and throughout the study, and for at least 4 months following the last study treatment.

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Female patients must have a negative serum beta-subunit of human chorionic gonadotropin (beta-hCG) pregnancy test (sensitivity of at least 25 mIU/mL) 28 days prior to registration on study and have a negative serum or urine (investigator's discretion under local regulations) β-hCG pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to the start of study treatment in the Treatment Period.

  * Note: the screening serum pregnancy test can be used as the test prior to the start of study treatment in the Treatment Period if it is performed within the 72-hour time frame)
* Male patients must agree to practice true abstinence from sexual intercourse or agree to the use of highly effective contraceptive methods (as described above) with non-pregnant female partners of child bearing potential at screening and throughout the course of the study and should avoid conception with their partners during the course of the study and for at least 4 months following the last study treatment.

  * Furthermore, the male subject must agree to use a condom while treated with ivosidenib and for at least 4 months following the last ivosidenib dose

Exclusion Criteria:

* Patients who are suspected or proven to have acute promyelocytic leukemia based on morphology, immunophenotype, molecular assay, or karyotype are not eligible
* Patients who have had prior therapy with ivosidenib are not eligible.

  * Note: prior treatment with other IDH inhibitors are allowed
* Patients who have immediate life-threatening, uncontrolled medical problem that would prevent treatment on a clinical trial per investigator's discretion are not eligible
* Patients who have significant active cardiac disease within 28 days prior to study registration, including New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 28 days prior to study registration are not eligible
* Patients who have prior history of malignancy, other than MDS, MPN, or AML are not eligible unless the subject has been free of the disease for >= 1 year prior to the start of study treatment. However, subjects with the following history/concurrent conditions are allowed:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Carcinoma in situ of the breast Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis clinical staging system)
* Patients who are known to have short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally are not eligible
* Patients who are taking the following sensitive CYP substrate medications that have a narrow therapeutic range are excluded from the study unless the subject can be transferred to other medications at least 5 half-lives or 14 days whichever is shorter prior to the start of study treatment: phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline, tizanidine (CYP1A2), CYP2C8, CYP3A4/5, and CYP2B6
* Patients who are known to be taking strong CYP3A4 inducers or sensitive CYP3A4 substrate medications that have a narrow therapeutic window are not eligible, unless they can be transferred to other medications within >= 5 half-lives prior to dosing or unless the medications can be properly monitored during the study
* Patients with an active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment) are not eligible
* Patients who have known or suspected hypersensitivity to any of the components of study therapy are not eligible
* Patient who has corrected QT (QTc) interval (Frederica's correction [QTcF]) >= 480 ms) at screening unless attributable to bundle branch block or pacemaker are not eligible. If prolonged QTc is attributed to medications the patient must be transferred to other medications and QTc corrected to selection parameters prior to enrollment
* Female patients who are pregnant or nursing are not eligible
* Patients who have any significant medical condition, laboratory abnormality, or psychiatric illness that the treating physician believes would prevent the subject from participating in the study are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | Up to day 42 of the first treatment cycle
  Will be assessed for a DLT per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose
  Will be assessed by the CTCAE version 5.0. Toxicity profiles will be summarized for toxicities of any grade, with rates of >= grade 3 toxicities also analyzed separately. Adverse events rates will be summarized and accompanied by 95% exact binomial confidence intervals.
Rates of complete remission (CR + complete remission with incomplete hematological recovery [CRi] + complete remission with incomplete platelet recovery [CRp]) | After induction on day 28 or upon count recovery, up to 1 year
  Patients that complete the induction cycle will be eligible for assessment
Progression free survival | At 1 year
  Will be estimated using Kaplan-Meier curves.
Overall survival | At 1 year
  Will be estimated using Kaplan-Meier curves.
Number of patients that receive hematopoietic stem cell transplant after induction treatment | Up to 1 year
  Patients that complete the induction cycle will be eligible for assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Shira N Dinner, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States